CLINICAL TRIAL: NCT06200051
Title: Multi-cancer Joint Screening and Early Diagnosis and Treatment Project
Brief Title: Multi-cancer Joint Screening and Early Diagnosis and Treatment Project Based on the Combination of Chinese Traditional and Western Medicine in Lanxi City
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Lanxi Hospital of Traditional Chinese Medicine (Other)
Collaborators: Zhejiang Chinese Medical University (Other Government); Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LX2023
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cancer Screening
Keywords: cancer screeing; traditional chinese medicine; risk; Lanxi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- High-risk group
  Interventions: Diagnostic Test: Prediction of high risk of cancer
- Moderate-risk group
  Interventions: Diagnostic Test: Prediction of high risk of cancer
- Low-risk group
  Interventions: Diagnostic Test: Prediction of high risk of cancer

INTERVENTIONS:
Diagnostic Test: Prediction of high risk of cancer — This initiative is aimed at comprehending the incidence rates of these four types of cancers, including lung cancer (LCA), liver cancer (LC), upper gastrointestinal cancer (UGIC), and CRC, to provide a theoretical foundation for the implementation of more practical and effective cancer screening strategies.

SUMMARY:
This study conducted a joint screening and early diagnosis and recommended treatment for LCA, LC, UGIC, and CRC among residents aged 45 to 74 in six townships of Lanxi City, Zhejiang Province. Residents who voluntarily participated and signed informed consent forms completed cancer risk assessment questionnaires and traditional Chinese medicine spleen deficiency (TCM-SD) investigations. The cancer risk assessment model established by the National Cancer Center was utilized to assess individual cancer risk scores. Simultaneously, blood samples (three tubes), one stool sample, and one urine sample were collected from each participant. Clinical screenings, including low-dose spiral CT, gastroscopy, colonoscopy, alpha-fetoprotein (AFP), and abdominal ultrasound, were performed for individuals identified as high-risk through the assessment.

DETAILED DESCRIPTION:
Screening Methods Population Selection for Screening: Utilizing a cluster sampling approach, one-fifth of the residents from six townships/districts were selected as the target population. Villages (communities) were organized and mobilized as units to central screening points. Work personnel were assigned to collaborate with local health institutions (community health service centers) to conduct a comprehensive survey of residents within their jurisdiction. The target population was registered and documented, and informed consent forms were obtained during this process.

Assessment of High-Risk Population: Utilizing a combination of questionnaire surveys and biological testing, the target population underwent risk assessment to identify individuals at high risk requiring clinical screening. Personnel administered the 'Cancer Risk Assessment Questionnaire (2022 edition)' and the 'Traditional Chinese Medicine Spleen Deficiency Questionnaire (TCM-SDQ)' to residents for a comprehensive assessment of multi-cancer disease risk. The questionnaire survey was conducted through face-to-face interviews by surveyors, with data entered into the 'Lanxi Multi-Cancer Joint Screening' data management platform. Ensuring residents fully understood the questionnaire content, maintaining the confidentiality of the survey, and ensuring the authenticity of the information were essential during the investigation. Additionally, on-site testing for Hepatitis B surface antigen (HBsAg), fecal occult blood test (FIT), and Helicobacter pylori (Hp) was carried out. Whole blood, feces, urine, and other samples were collected on the same day for biological testing.

Clinical Screening: For individuals identified as high-risk for cancer by the risk assessment system, they were informed of their cancer risk and organized to undergo specified clinical screenings at designated hospitals. The clinical screenings included low-dose CT (LDCT) for the lungs, upper gastrointestinal endoscopy with targeted indicated pathological biopsy, colonoscopy with targeted indicated pathological biopsy, AFP detection and liver ultrasound, molybdenum target, and ultrasound, among others. The screening protocols for the five common cancers (lung, upper gastrointestinal, colorectal, liver) followed the 'Urban Cancer Screening and Early Diagnosis and Treatment Project Technical Plan (2022 edition).' Results from clinical screenings were systematically recorded in the 'Lanxi City Multicancer Integrated Screening' data management platform.

Population Follow-up: For individuals identified as high-risk in the past and requiring follow-up, notifications were sent through the information platform. Project unit staff, following the screening tasks, collected information on the diagnosis and treatment of the follow-up subjects. Follow-up activities were conducted actively and passively, employing methods such as direct face-to-face visits, telephone interviews, self-administered questionnaires, regular physical examinations, environmental and disease monitoring, and collection of attendance records from hospitals and workplaces. The active follow-up targeted individuals with positive findings of various cancers detected through clinical examinations in the past (specific criteria outlined in the 'Urban Cancer Screening Early Diagnosis and Treatment Project Follow-up Plan'). Active follow-up involved undergoing clinical examinations again and collecting follow-up information. Among them, those undergoing clinical examinations were included in the annual completion volume. Follow-up information included detailed information on diagnosis and treatment. For de-ceased individuals, specific death information (including time and cause of death, etc.) needed to be obtained. Passive follow-up involved matching the project participants with the local cancer registry and cause-of-death monitoring database to supplement information on cancer incidence and death among project participants.

ELIGIBILITY:
Inclusion Criteria:

* The survey focused on residents aged 45 to 74 years, based on their permanent residency status (The date of birth on the ID card shall prevail).
* All participants possessed full legal capacity and voluntarily signed informed consent forms.

Exclusion Criteria:

* Individuals who had moved out, long-term absence, or had household separation were excluded. The screening participants were further confirmed to meet the eligibility criteria after excluding those with poor compliance, already diagnosed with tumors, or having severe heart, brain, lung diseases, or renal dysfunction.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Utilizing a cluster sampling approach, one-fifth of the residents from six town-ships/districts were selected as the target population. Villages (communities) were organized and mobilized as units to central screening points. Work personnel were assigned to collaborate with local health institutions (community health service centers) to conduct a comprehensive survey of residents within their jurisdiction. The target population was registered and documented, and informed consent forms were obtained during this process.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
program coverage rate | 2024.01-2026.12
  percentage of people guided by navigators
screening participation rate | 2024.01-2026.12
  Screening participation rate (%) is determined by the number of clinical screening cases divided by the number of cases identified as high-risk, multiplied by 100%.
high-risk rate | 2024.01-2026.12
  The high-risk rate (%) is calculated as the high-risk individuals identified divided by the total number of participants in the assessment, multiplied by 100%.
Positive lesion detection rate | 2024.01-2026.12
  Positive lesion detection rate is calculated as the number of clinically detected positive lesions divided by the total number of screened cases, multiplied by 100%.
Detection rate | 2024.01-2026.12
  Detection rate is computed as the number of confirmed cancer cases divided by the total number of screened cases, multiplied by 100%.

SECONDARY OUTCOMES:
Risk factor investigation | 2024.01-2026.12
  According to the findings of CRAQ and TCM-SDQ, the risk factors were investigated, including dietary habits, living environment, lifestyle, medical history, family history of malignancies, past medication history, female physiology, reproductive history, and pri-marily TCM-SD symptoms
Awareness rate of cancer prevention and treatment among residents | 2024.01-2026.12
  To objectively assess the level of cancer prevention and control knowledge among resi-conduct a survey based on the Cancer Prevention and Con-trol Core Knowledge Awareness Survey Scale released by the NCC.
Cost effectiveness analysis | 2024.01-2026.12
  In order to estimate the cost-effectiveness of the implementation of such a program, mar-ginal costs, with encryption on the actual cost, observed during the installation, as well as a projection on a routine cost will be taken into account.
5-year cancer survival rate | 2024.01-2029.12
  We will employ a combination of proactive and passive follow-ups, along with linkage to the city's population database and mortality database, to calculate the five-year survival rates for patients with four types of cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Jing Xiao, Lanxi, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No